CLINICAL TRIAL: NCT04344964
Title: Endoscopy-related Phone Consultation During the COVID-19 Outbreak: Impact on Attendance and Patient/Consultant Perspectives From a Tertiary Australian Hospital
Brief Title: Endoscopy-related Phone Consultation During the COVID-19 Outbreak
Status: Completed | Type: Observational
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Leonardo Zorron Cheng Tao Pu, Endoscopy Fellow, Austin Health
Other Study IDs: 38839
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Colon Polyp; Colon Disease; Reflux, Gastroesophageal; Varices, Esophageal
MeSH Terms: conditions — Colonic Polyps; Colonic Diseases; Gastroesophageal Reflux; Esophageal and Gastric Varices

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phone consult group: Information collected prospectively on FTA patients and questionnaire (satisfaction)
  Interventions: Other: None - NA
- Face-to-face consult group: Information collected retrospectively on FTA patients
  Interventions: Other: None - NA

INTERVENTIONS:
Other: None - NA — Observational study

SUMMARY:
The aim of this study is to evaluate patient and consultant experiences with phone consultations for endoscopy-related outpatient appointments during the COVID-19 outbreak.

DETAILED DESCRIPTION:
Telephone consultations as a method for telehealth do not provide visual cues and limit interpretation of visual signs such as visualization of skin lesions. However, the need of such feedback is almost non-existent for endoscopy-related consultations as their purpose is focused. The main foci of endoscopy-related outpatient clinics are two: 1 - inform and consent the patient for an endoscopic procedure that is to be done in the near future; 2 - explain the results of a recent procedure already performed and which has a copy provided to the patient. Therefore, phone consultations might be a good fit for endoscopy-related outpatient clinics. The practicalities and indications for the use of phone consults has been described by van Galen & Car (2018) and fit the above description.

Patients will be invited to participate only after the consultation have been finalised and all questions regarding the endoscopic procedure to be done/that was done have been clarified. Patients and consultants will fill questionnaires to evaluate the phone consultation.

The primary outcome will the the comparison of "failed to attend" (FTA) occurrences compared to a similar period of the past year. Secondary outcomes will be patients' and consultants' satisfaction with the phone consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patients booked for an outpatient consultation in the Post-Endoscopy clinic or Advanced Endoscopy clinic
* Consultation determined to be held over the phone as per preventive measures due to the COVID-19 outbreak
* Age > 18 years
* Ability to give informed consent

Exclusion Criteria:

* Phone consultation done with a relative as per patient's preference or inability to talk over the phone
* Patient that is deemed as confused/not able to understand
* Unwilling/unable to participate in the post-consultation survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that have been submitted or were ordered any endoscopic procedure (e.g. capsule endoscopy, enteroscopy, endoscopic mucosal resection) within Austin Health - Victoria - Australia.
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Failed to attend patients | 2 months
  percentage of patients that did not answer phone calls (at least 3 calls) or with documented FTA for the retrospective group.

SECONDARY OUTCOMES:
Patient satisfaction with the phone consult | 2 months
  Assessed through an online/hardcopy questionnaire based on previous studies on telehealth (adapted from Barsom et al. 2020 - MSF and PAT-VC questionnaires). These are mostly Likert-scale response mode statements.
Consultant satisfaction with the phone consult | 2 months
  Assessed through an online/hardcopy questionnaire based on previous studies on telehealth (adapted from Barsom et al. 2020). These are mostly Likert-scale response mode statements.

CONTACTS AND LOCATIONS:
Overall Officials: Sujievvan Chandran, MD, Principal Investigator — Consultant Gastroenterologist
Locations (1):
- Austin Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
For ethical purposes as per the approval of this study as a quality improvement study (and hence exempted of formal HREC evaluation). Data should be shared outside Austin Health only through grouped data in conferences and journal papers.

REFERENCES:
- [Background] Barsom EZ, Jansen M, Tanis PJ, van de Ven AWH, Blusse van Oud-Alblas M, Buskens CJ, Bemelman WA, Schijven MP. Video consultation during follow up care: effect on quality of care and patient- and provider attitude in patients with colorectal cancer. Surg Endosc. 2021 Mar;35(3):1278-1287. doi: 10.1007/s00464-020-07499-3. Epub 2020 Mar 20. PMID 32198552
- [Background] van Galen LS, Car J. Telephone consultations. BMJ. 2018 Mar 29;360:k1047. doi: 10.1136/bmj.k1047. No abstract available. PMID 29599197